CLINICAL TRIAL: NCT00569894
Title: A Post Marketing Evaluation of the Safety of FluMist in Children 24-59 Months of Age in a Managed Care Setting
Brief Title: A Post Marking Study to Evaluate the Safety of FluMist in Children
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Medical Monitor, MedImmune, LLC
Other Study IDs: MI-MA162
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2: TIV
  Interventions: Biological: TIV (Injection)
- 1: FluMist
  Interventions: Biological: FLuMist
- 3: Unvaccinated
  Interventions: Other: Unvaccinated Control

INTERVENTIONS:
Biological: FLuMist — One or two vaccinations with FluMist depending on prior vaccination status.
  Groups: 1
Biological: TIV (Injection) — One or two injections of TIV depending on previous status.
  Groups: 2
Other: Unvaccinated Control — no vaccine
  Groups: 3

SUMMARY:
To assess the safety of FluMist vaccination

DETAILED DESCRIPTION:
* To assess the safety of FluMist vaccination Rates of medically attended events in FluMist recipients, including serious adverse events (SAEs), anaphylaxis , urticaria, asthma, wheezing, pre-specified grouped diagnoses, and rare events potentially related to wild-type influenza, will be compared to rates in multiple non-randomized control groups.
* To assess the safety of annual FluMist re-vaccination [Rates of MAEs in the subset of children who receive FluMist in ≥2 consecutive years will be compared to rates in first-time vaccinees during the same season.]
* To assess the safety of FluMist vaccination in children previously vaccinated with trivalent inactivated influenza vaccine (TIV) [Rates of MAEs in the subset of children who received one or more prior TIV vaccinations will be compared to rates in children who did not receive prior TIV.]

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age: born within the same calendar quarter as the reference FluMist vaccinee.

Exclusion Criteria:

* Children who have evidence of medical conditions that put them at high risk for complications of influenza (e.g., chronic cardiovascular and pulmonary disease) will be excluded from this control group.

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The populations to be assessed are FluMist recipients, TIV recipient controls, and unvaccinated controls.
  Members of the Kaiser Permanente Health Care Plan may be included in this study as part of routine care at their participating health centers within the Kaiser Permanente health maintenance organization (HMO) of Northern California.
Sampling Method: Probability Sample
Enrollment: 29296 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Assess Medically Attended Events(MAEs)of anaphylaxis,urticaria, asthma,wheezing,pre-specified grouped diagnoses,and rare events related to wild-type influenza,MAEs-qualify as SAEs,in:emergency department,clinic,and hospital setting. | 1, 3, 21, or 42 days post dose; 6 months post dose; entire study period)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Toback, M.D., Study Director — MedImmune LLC
Locations (1):
- Research Site, Oakland, California, United States